CLINICAL TRIAL: NCT06733493
Title: Integrated Psychosocial Care in Intensive Care: Piloting of an Innovative Care Approach (IPS Pilot) - Study Protocol for a Pilot Randomized Controlled Trial
Brief Title: Study Protocol for a Pilot Randomized Controlled Trial of a Psychosocial Care Intervention in Intensive Care
Acronym: IPS-Pilot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harald Gündel (Other)
Collaborators: Institute of Social Medicine and Health Systems Research, University Hospital Magdeburg (Unknown); University Hospital Berlin Charite (Unknown); Magdeburg University Hospital, Germany (Unknown)
Responsible Party: Sponsor-Investigator, Harald Gündel, Prof. Harald Gündel, University Hospital Ulm
Organization: University Hospital Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01VSF22020; 01VSF22020 (Other Grant/Funding Number: German Federal Joint Committee (G-BA))
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Psychosocial Intervention; Intensive Care Units (ICUs); Psychosocial Health
Keywords: health services research; psychosocial intervention; health personnel; INTENSIVE CARE UNIT; Critical Care

STUDY DESIGN:
Intervention Model Description: Multi-center study on 3 sites and 8 ICU wards, with cluster-randomization of intervention (n=4) and control wards (n=4).
  Data-collection in a mixed design:
  * Between-subject factor: Affiliation to intervention or control ICU ward
  * Between-subject factor: Affiliation to the group of healthcare professionals, relatives or patients
  * Within-subject factor: Time of data collection (baseline or follow-up)
  * Healthcare professionals: baseline (first 6 weeks of treatment) and follow-up (last 6 weeks of treatment)
  * Relatives: baseline (during treatment of their patient in the ICU and up to 4 weeks after), follow-up (4 months after completing baseline)
  * Patients: No baseline data-collection since this would produce a biased sample (only mildly impaired ICU patients), follow-up (4 months after ICU stay)
Who Masked: Participant
Masking Description: Participating Healthcare-professionals can not be fully masked, since they are aware of the new team member in form of a ward psychologist (intervention) or aware that a ward psychologist was employed in another ward (control). Yet they are not aware about key efficacy components of the intervention (as the team integration, mere presence, ...)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IPS-Intervention Group (Experimental): Implementation of a trained ward psychologist for 12 months, supporting patients, relatives and staff according to the IPS-intervention manual
- Control Group: Standard Care (No Intervention): No intervention will be admitted. ICU wards receive the usual care, e.g. consiliary psychological service, optional consultation for staff

INTERVENTIONS:
Behavioral: integrated psychosocial care — Employment of a psychologist in psychotherapeutic training as a member of the multiprofessional team at the ICU ward for the duration of one year. Tasks: Psychosocial Support for staff, patients and their relatives.
  Other Names: IPS-intervention; ward psychologist; IPS study therapist; IPS study psychologist

SUMMARY:
This Pilot-RCT is part of a feasibility study that aims to learn if the IPS-psychosocial care intervention and an RCT on its efficacy are feasible in patients, relatives and staff on icu wards. The Pilot-RCT will examine outcomes, that might indicate an improvement in psychosocial safety climate and other health- and wellbeing-related measures due to the administration of the intervention that is described in the following. The main question the Pilot-RCT aims to answer is:

Is there evidence that the IPS intervention improves the psychosocial safety climate and other components of psychosocial well-being in ICU teams, patients and their relatives?

Researchers will compare four intervention groups (icu wards with implementation of the IPS-Intervention) with four control groups (icu wards with regular supply of psychosocial care) to see if the comparison of two groups in this RCT is feasible.

The IPS-Intervention consists of a ward psychologist who works as part of the ICU team and takes care of the staff, patients and relatives in accordance to the intervention manual that was developed in a prior phase of this project.

ELIGIBILITY:
Inclusion Criteria:

* Affiliation to one of the 8 participating ICU wards during the duration of the study, either by: occupation as a healthcare professional, admission as a patient, relation to an admitted patient

Exclusion Criteria:

* Age under 18 years old
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Psychosocial Safety Climate | Baseline (first 6 weeks of treatment) and Follow-Up (last 6 weeks of treatment)
  Psychosocial Safety Climate as perceived by ICU staff in the experimental and control group, measured with the German version of the Psychosocial Safety Climate (PSC-4) scale (Formazin, Ertel, Kersten, & Nübling, 2022). 4 items (eg. "Senior management shows support for stress prevention through involvement and commitment") ranked on a 5-point Likert scale (1 = Strongly disagree, 5 = Strongly agree). A higher sum score of the 4 items (Min = 4, Max = 20) indicates a more positive psychosocial safety climate
Intention to leave | Baseline (first 6 weeks of treatment) and Follow-Up (last 6 weeks of treatment)
  Healthcare Professionals' Intention to leave their workplace, profession or reduce their working time, measured with the questions from the Nurses Early Exit (NEXT) study (Simon, Tackenberg, Hasselhorn, Kümmerling, Büscher, & Müller, 2005). 3 items ranked on a 5-point Likert-scale. A higher sum score (Min=3, Max=15) indicates a higher turnover intention.
Perceived Wellbeing | Healthcare Professionals: Baseline and Follow-Up; Relatives: Baseline and Follow-Up; Patients: 4 months after ICU stay
  Healthcare professionals', patients', and relatives' perceived well-being, measured with the german version of the WHO-5 (World Health Organization-Five) wellbeing index (Brähler, Mühlan, Albani, & Schmidt, 2005). 5 items rated on a 6-point Likert scale ranging from 0 (At no time) to 5 (All of the time). Higher overall sumscores (Min=0, Max=25) indicate better well-being.
Health-related quality of life | Healthcare Professionals: Baseline and Follow-Up; Relatives: Baseline and Follow-Up; Patients: 4 months after ICU stay
  Healthcare professionals', patients', and relatives' perceived health-related quality of life, measured with the german version of the Short-Form Health-Related Survey (SF-12, Drixler, Morfeld, Glaesmer, Brähler, Wirtz, 2020). 12 items with a mixed response format (2-6 options) that can be assigned to the Physical Component Summary (PCS) and Mental Component Summary (MCS). PCS and MCS are standardized (Mean = 50, SD = 10). Higher scores indicate better physical or mental health-related quality of life.
Perceived Stress | Healthcare Professionals: Baseline (first 6 weeks of treatment) and Follow-Up (last 6 weeks of treatment); Relatives: Baseline (during first 8 months of treatment, individually: during or up to 4 weeks after ICU admission), Follow-Up: 4 months after Base
  Healthcare professionals', patients' and relatives' perception of stress, measured with the german version of the Perceived Stress Scale (PSS-10, Klein, Brähler, Dreier, Reinecke, Müller, Schmutzer, Wölfling, & Beutel, 2016). 10 items that are rated on a 5-point Likert scale from 0 (Never) to 4 (Very often). Higher total scores (Min=0, Max=40) reflect higher perceived stress.
Depression / Anxiety | Healthcare Professionals: Baseline and Follow-Up; Relatives: Baseline and Follow-Up; Patients: 4 months after ICU stay
  Healthcare professionals', patients', and relatives' perceived depressive and anxiety symptoms, measured with the german version of the patient health questionnaire (PHQ-4, Löwe, 2015). 4 items rated on a 4-point Likert scale from 0 (Not at all) to 3 (Nearly every day). Higher total scores (Min=0, Max=12) indicate more severe psychological distress.
Work-related consequences of strain | Baseline (first 6 weeks of treatment) and Follow-Up (last 6 weeks of treatment)
  Emotional and cognitive irritation as perceived by ICU staff in the experimental and control group, measured with the irritation scale to measure consequencey of work-related strain (Mohr, Rigotti, & Müller, 2007). 8 items rated on a 7-point Likert scale from 1 (Strongly disagree) to 7 (Strongly agree). Higher total scores for the overall irritation scale (Min=8, Max=56), Emotional Irritation subscale (5 items, Min=5, Max=35) and Cognitive Irritation (3 items, Min=3, Max=21) indicate higher levels of irritation.
Self-efficacy, optimism and pessimism | Healthcare Professionals: Baseline and Follow-Up; Relatives: Baseline and Follow-Up; Patients: 4 months after ICU stay
  Healthcare professionals', patients', and relatives' perceived self-efficacy, optimism and pessimism measured with the german self-efficacy, optimism and pessimism questionnaire (SWOP-K9, Scholler, Fliege, & Klapp, 1999). 9 items rated on a 4-point scale from 1 (Does not apply at all) to 4 (Applies completely) and are divided into the subscales self-efficacy, optimism and pessimism. Higher subscale means (Min=1, Max=4) for self-efficacy and optimism indicate better psychological resources; higher pessimism subscale means indicate worse outcomes.
Team cohesion at work | Baseline (first 6 weeks of treatment) and Follow-Up (last 6 weeks of treatment)
  Team cohesion in the ICU as perceived by ICU staff in the experimental and control group, measured with the Erlangen Team Cohesion at work scale (ETC, Lieb, Erim, & Morawa, 2024). 13 items rated on a 5-point Likert scale (1 = Strongly disagree, 5 = Strongly agree) and can be divided into the subsales Collegial Solidarity and Unity and Problem Management. A higher overall sum score (Min=13, Max=65) or higher subscale means (Min=1, Max=5) indicate stronger team cohesion.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Gündel, Prof. Dr. med., Principal Investigator — Clinic of Psychosomatic Medicine and Psychotherapy, University Hospital Ulm,
Locations (4):
- Germany (4):
  - Clinic of Psychosomatic Medicine and Psychotherapy, University Hospital Ulm, Ulm, Baden-Wurttemberg
  - Psychosomatic Medicine and Psychosomatic Therapy, Medical Faculty University Hospital Magdeburg, Magdeburg, Saxony-Anhalt
  - Institute of Social Medicine and Health Systems Research (ISMHSR), Magdeburg, Saxony-Anhalt
  - Medical Clinic - Department of Psychosomatic Medicine of the Charité, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nickel SF, Korger S, Schindler W, Heytens H, Krieg G, Drewitz KP, Schurmann K, Schossow L, Gehrig J, Binnebose M, Hirning C, Honig K, Niessen RK, Kirschbaum J, Erdur L, Peter S, Junne F, Rose M, Apfelbacher C, Gundel H. Integrated Psychosocial Care in Intensive Care (IPS-Pilot): Protocol for the Systematic, Multimethod Development of a Complex Intervention (Phase A). JMIR Res Protoc. 2025 Jun 6;14:e65682. doi: 10.2196/65682. PMID 40479723
- See also: Registry of the study with the funder — https://innovationsfonds.g-ba.de/projekte/versorgungsforschung/ips-pilot-integrierte-psychosoziale-versorgung-in-der-intensivmedizin-partizipative-entwicklung-und-pilotierung-eines-innovativen-versorgungsansatzes.530
- See also: Project Registry at OSF — https://osf.io/vfxjk/